CLINICAL TRIAL: NCT04611464
Title: Pain and Functional Outcomes With Misoprostol Treatment for Lumbar Spinal Stenosis
Brief Title: Misoprostol for Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thiru Annaswamy, Professor, PM&R, Principal Investigator, Staff Physician, Dallas VA Medical Center
Other Study IDs: 19-006
Record Dates: First submitted 2020-10-09; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Lumbar Spinal Stenosis; Low Back Pain
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain | interventions — Misoprostol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Single-group cross-sectional cohort: Patients who have previously received off-label prescriptions of misoprostol for lumbar spinal stenosis for any duration and who are willing to provide verbal and informed consent.
  Once enrolled, patients will complete the Swiss Lumbar Spinal Stenosis Questionnaire (SSSQ) as well as the Oswestry Disability Index (ODI). The SSSQ will elicit patients' responses specifically related to their usage of misoprostol for lumbar spinal stenosis.
  Then their walking tolerance will be assessed by having them walk along a measured walkway of up to 500 feet to determine the onset of their neurogenic claudication symptoms at a certain distance, their claudication distance.
  Prescription information on dosage and frequency of misoprostol use, and any reported side effects with use of this medication, and any cessation or stoppage of use of this medication will all be recorded.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Misoprostol is a PGE1 analog

SUMMARY:
This single-group cross-sectional cohort study will enroll approximately 25 patients at the North Texas VA Health Care System (VANTHCS) who have previously received off-label prescriptions of misoprostol for lumbar spinal stenosis for any duration and who are willing to provide verbal and informed consent. Patients will answer a questionnaire regarding pain and functional improvement especially in reference to misoprostol treatment. Patients will also be selected to have their walking tolerance (claudication distance) measured in an outpatient clinic setting to determine the severity of their lumbar spinal stenosis symptoms after having received misoprostol.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is clinically described as a neurogenic claudication that is associated with increased mechanical compression on the spinal nerve roots as well as potential compromise of the vascular supply of the spinal nerve roots. This compression typically leads to symptoms of lumbar pseudoclaudication, which include pain, paresthesias, and discomfort in the lower extremities, commonly exacerbated by walking. Broadly speaking, this compression can be the result of a degenerative narrowing of the spinal or nerve root canals. While spinal stenosis is typically considered idiopathic, causes can also include malignancy, injury, and chronic inflammation. It is often debilitating to patients and can lead to a wide variety of negative health outcomes (pre-operative lower levels of function, psychological distress, high self-reported disability scores and operative risks of surgical correction) related to attempted surgical correction of lumbar spinal stenosis. Spinal stenosis continues to be a leading indication for spine surgery in adults older than 65 years old. Furthermore, estimated total Medicare costs for surgeries treating lumbar spinal stenosis amounted to over $1.65 billion for 37,598 individual operations.

Physiologically, the venous blood flow in the lumbar spinal region is disproportionately affected by pressure gradients generated secondary to normal movement and pathologic constriction. Studies have found that patients diagnosed with lumbar spinal stenosis with intermittent claudication, while walking on a treadmill, experienced larger amounts of vascular congestion which resolved with sitting. This was measured with a myeloscope in the intrathecal space.

The current vascular pathologic mechanism of the symptomatic effects of lumbar spinal stenosis is thought to be a consequence of constriction leading to increasing vascular congestion and inflammation. Authors first described the effect of constriction on vascular flow through a post mortem study of a patient with chronic lumbar spinal stenosis at L4-L5. Most significantly, they found that venous supply proximal to constriction in fact showed reduced and collapsed veins with gross congestion proximal to the lesion. Further investigation found that venous congestion led to increased inflammatory markers in nerves with atrophy, Wallerian degeneration, and perineural fibrosis in more severe patients. Most importantly, these pathologic changes were associated with vascular changes in the absence of direct nerve root compression at these sites. This venous congestion is a potential target for therapy.

There has been previous work done with medications that are PGE1 analogs such as limaprost and lipo-PGE1. PGE1 analogs hypothetically treat the above lumbar spinal stenosis pathology by improving blood flow to nerve roots through vasodilatory and antiplatelet aggregation effects. However, misoprostol (PGE1 analog) has not been thoroughly evaluated as a possible treatment for symptoms of lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Previous diagnosis of lumbar spinal stenosis, mild-severe lumbar central canal stenosis identified by MRI or CT scan.
* Symptoms:

  * Lower extremity symptoms consistent with neurogenic claudication.
  * Pain, weakness &/or numbness triggered by standing or walking, and relieved by sitting.
* Must be able to read English and complete questionnaire.
* Was prescribed Misoprostol specifically for lumbar spinal stenosis.

Exclusion Criteria:

* Cognitive impairment that renders the patient unable to give informed consent or provide accurate data
* Clinical co-morbidities that could interfere with the collection of data concerning pain and function
* Severe vascular, pulmonary, or coronary artery disease that limits ambulation including recent myocardial infarction (within 6 months)
* Spinal instability requiring surgical fusion
* Severe osteoporosis as defined by multiple compression fractures or a fracture at the same level as the stenosis
* Metastatic cancer
* Excessive alcohol consumption or evidence of non-prescribed or illegal drug use
* Pregnancy
* Concordant pain with internal rotation of the hip (or known hip joint pathology)
* Active local or systemic infection
* Previous lumbar spine surgery
* Prisoners
* Use of misoprostol for any other indication then lumbar spinal stenosis
* Rheumatological disorders such as rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single-group cross-sectional cohort study will enroll approximately 25 patients at the North Texas VA Health Care System (VANTHCS) who have previously received off-label prescriptions of misoprostol for lumbar spinal stenosis for any duration and who are willing to provide verbal and informed consent.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Swiss Lumbar Spinal Stenosis Questionnaire(SSSQ) | Once at baseline, after they have been treated with Misoprostol; SSSQ has not been collected previously
  The SSSQ quantifies severity of symptoms, physical function characteristics, and patient's satisfaction after treatment.
Oswestry Disability Index (ODI) | Change from baseline, after they have been treated with Misoprostol
  The ODI quantifies disability dues to lumbar spinal stenosis symptoms
Claudication Distance Assessment | Change from baseline, after they have been treated with Misoprostol
  Measure walking tolerance to determine the severity of their lumbar spinal stenosis symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States